CLINICAL TRIAL: NCT02282020
Title: A Phase III, Open Label, Randomised, Controlled, Multi-centre Study to Assess the Efficacy and Safety of Olaparib Monotherapy Versus Physician's Choice Single Agent Chemotherapy in the Treatment of Platinum Sensitive Relapsed Ovarian Cancer in Patients Carrying Germline BRCA1/2 Mutations.
Brief Title: Olaparib Treatment in Relapsed Germline Breast Cancer Susceptibility Gene (BRCA) Mutated Ovarian Cancer Patients Who Have Progressed at Least 6 Months After Last Platinum Treatment and Have Received at Least 2 Prior Platinum Treatments
Acronym: SOLO3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Myriad Genetic Laboratories, Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: D0816C00010
Expanded Access: NCT03079687 (Approved for marketing)
Record Dates: First submitted 2014-10-20; First posted 2014-11-04 (Estimated); Results first posted 2019-12-02 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Relapsed Ovarian Cancer, BRCA Mutation, Platinum Sensitivity
Keywords: BRCA, ovarian, platinum, chemotherapy,
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1/OLAPARIB (Experimental): olaparib 300mg oral tablets; twice daily
  Interventions: Drug: OLAPARIB
- 2/CHEMOTHERAPY (Active Comparator): Physician's choice single agent chemotherapy
  Interventions: Drug: Single agent chemotherapy

INTERVENTIONS:
Drug: OLAPARIB — 300 mg olaparib tablets taken orally twice daily. All patients should continue to receive study treatment until objective radiological disease progression as per RECIST 1.1 as assessed by the investigator or the patient experiences unacceptable toxicity or they meet any other discontinuation criteria.
  Arms: 1/OLAPARIB
Drug: Single agent chemotherapy — Treatment of relapsed disease with single agent chemotherapy based on physician's choice of weekly paclitaxel, topotecan, pegylated liposomal doxorubicin, or gemcitabine. All patients should continue to receive study treatment until objective radiological disease progression as per RECIST 1.1 as assessed by the investigator or the patient experiences unacceptable toxicity or they meet any other discontinuation criteria
  Arms: 2/CHEMOTHERAPY

SUMMARY:
Comparison of olaparib vs. physician's choice of single agent standard of care non-platinum based chemotherapy in patients with germline Breast Cancer susceptibility gene (gBRCA) mutated ovarian cancer who have progressed at least 6 months after the last platinum based chemotherapy. Patient should have received at least 2 prior lines of platinum based chemotherapy. The aim of the study is to assess the efficacy and safety of olaparib tablets.

DETAILED DESCRIPTION:
This open label, randomised, controlled, multi-centre study will assess the efficacy and safety of single agent olaparib vs. standard of care, based on physician's choice of single agent chemotherapy ( i.e paclitaxel, or topotecan, or pegylated liposomal doxorubicin, or gemcitabine) in platinum sensitive or partially platinum sensitive relapsed ovarian cancer patients who carry germline deleterious or suspected deleterious BRCA mutation and who have received at least 2 prior lines of platinum based chemotherapy. Patients are eligible to undergo BRCA testing even if they have not yet had recurrence or progression of disease >6 months (>/=183 days) after completion of their last platinum therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years of age
* Patients with histologically diagnosed relapsed high grade serous ovarian cancer (including primary peritoneal and/or fallopian tube cancer) or high grade endometrioid cancer. Patients are eligible to undergo BRCA testing even if they have not yet had recurrence or progression of disease >6 months (>/=183 days) after completion of their last platinum therapy.
* Documented germline mutation in Breast Cancer susceptibility genes: BRCA1 and/or BRCA2 that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function)
* At least one lesion that can be accurately assessed at baseline by CT/MRI and is suitable for repeated assessment.
* Patients must have received at least 2 prior platinum based lines of chemotherapy - Patients must be partially platinum sensitive or platinum sensitive
* Patients must be suitable to start treatment with single agent chemotherapy based on physician's choice
* Patients must have normal organ and bone marrow function measured within 28 days of randomisation,
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must have a life expectancy ≥ 16 weeks
* Formalin fixed, paraffin embedded tumour sample from the primary or recurrent cancer must be available for central testing.

Exclusion Criteria:

* BRCA 1 and/or BRCA2 mutations that are considered to be non detrimental
* Exposure to any investigational product within 30 days or 5 half lives (whichever is longer) prior to randomisation
* Any previous treatment with a Polyadenosine 5'diphosphoribose polymerisation (PARP) inhibitor, including olaparib.
* Patients who have platinum resistant or refractory disease
* Patients receiving any systemic chemotherapy within 3 weeks prior to first dose of study treatment
* Previous single agent exposure to the selected chemotherapy regimen for randomisation. - Prior malignancy in the last 5 years, unless curatively treated and recurrence free (few exceptions apply).

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2015-02-06 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2022-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Penson, Associate Prof. of Medicine, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (77):
- United States (22):
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Sacramento, California
  - Research Site, San Francisco, California
  - Research Site, Aurora, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Hartford, Connecticut
  - Research Site, Fort Gordon, Georgia
  - Research Site, Covington, Louisiana
  - Research Site, Towson, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Albany, New York
  - Research Site, Mineola, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Springfield, Oregon
  - Research Site, Abington, Pennsylvania
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Bedford, Texas
  - Research Site, Houston, Texas
  - Research Site, Milwaukee, Wisconsin
- Argentina (6):
  - Research Site, Berazategui
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, San Miguel de Tucumán
- Belgium (2):
  - Research Site, Ghent
  - Research Site, Leuven
- Brazil (6):
  - Research Site, Ijuí
  - Research Site, Passo Fundo
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Czechia (4):
  - Research Site, Hradec Králové
  - Research Site, Ostrava-Poruba
  - Research Site, Prague
  - Research Site, Zlín
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Miskolc
- Israel (10):
  - Research Site, Afula
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Rehovot
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
  - Research Site, Ẕerifin
- Italy (5):
  - Research Site, Meldola
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Roma
- Mexico (2):
  - Research Site, México
  - Research Site, Oaxaca City
- Poland (7):
  - Research Site, Gdansk
  - Research Site, Grzepnica
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Warsaw
- South Korea (2):
  - Research Site, Goyang-si
  - Research Site, Seoul
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Girona
  - Research Site, Granada
  - Research Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Scambia G, Villalobos Valencia R, Colombo N, Cibula D, Leath CA 3rd, Bidzinski M, Kim JW, Nam JH, Madry R, Hernandez C, Mora PAR, Ryu SY, Ah-See ML, Lowe ES, Lukashchuk N, Carter D, Penson RT. Olaparib as Treatment Versus Nonplatinum Chemotherapy in Patients With Platinum-Sensitive Relapsed Ovarian Cancer: Phase III SOLO3 Study Final Overall Survival Results. J Clin Oncol. 2025 Apr 20;43(12):1408-1416. doi: 10.1200/JCO.24.00933. Epub 2024 Dec 12. PMID 39668137
- [Derived] Paulino E, Melo AC. SOLO 3 Trial: How Do the Results Fit in With Current Evidence? J Clin Oncol. 2020 Aug 10;38(23):2697-2698. doi: 10.1200/JCO.20.00576. Epub 2020 Jun 12. No abstract available. PMID 32530768
- [Derived] Penson RT, Lowe ES. Reply to E. Paulino et al. J Clin Oncol. 2020 Aug 10;38(23):2698. doi: 10.1200/JCO.20.01235. Epub 2020 Jun 12. No abstract available. PMID 32530766
- [Derived] Penson RT, Valencia RV, Cibula D, Colombo N, Leath CA 3rd, Bidzinski M, Kim JW, Nam JH, Madry R, Hernandez C, Mora PAR, Ryu SY, Milenkova T, Lowe ES, Barker L, Scambia G. Olaparib Versus Nonplatinum Chemotherapy in Patients With Platinum-Sensitive Relapsed Ovarian Cancer and a Germline BRCA1/2 Mutation (SOLO3): A Randomized Phase III Trial. J Clin Oncol. 2020 Apr 10;38(11):1164-1174. doi: 10.1200/JCO.19.02745. Epub 2020 Feb 19. PMID 32073956
- See also: AstraZeneca Cancer Study Locator Service Phone 677 400 4656 Email astrazeneca@emergingmed.com — http://emergingmed.com/networks/AstraZeneca
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00010&attachmentIdentifier=041c3c95-2c81-475b-ae11-1769903a7112&fileName=20190614_SOLO-3_d0816c00010_Protocol_Amendment-v4_20Dec17_Final_Redacted_(1).pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00010&attachmentIdentifier=4ef96d32-3bc9-474b-8bcf-0c6fd80190aa&fileName=20190614_AZ_SOLO-3_Statistical_Analysis_Plan_v4_30-Oct-2018_Final_Redacted_(1).pdf&versionIdentifier=
- See also: CSR Synopsis addendum — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00010&attachmentIdentifier=0e755241-5571-4243-b9f4-92b1001d85b3&fileName=d0816c00010-add2-CSRsynopsis-redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 678 patients were screened (gave informed consent) at 94 centres in 13 countries. Of the 678 patients screened, 266 patients were randomised from 78 sites in 13 countries worldwide.
  A wash-out period of up to 5 weeks was required for participants who have previously taken potent inhibitors or CYP3A4/5 inducers.
Pre-assignment Details: Participants were randomized in a 2:1 ratio between olaparib and single agent chemotherapy. Of the 266 patients randomised, 178 patients were in the olaparib arm and 88 in the chemotherapy arm.
Groups:
- Olaparib 300mg BID: Participants received olaparib twice daily as a 300 mg tablet.
- Single Agent Chemotherapy: Participants received physician's choice of chemotherapy, out of weekly paclitaxel, topotecan, pegylated liposomal doxorubicin, or gemcitabine.
Period: Overall Study
Arm/Group | Olaparib 300mg BID | Single Agent Chemotherapy
Started | 178 | 88
Received Treatment | 178 | 76
Completed (Ongoing study treatment at time of analysis DCO: 16 April 2021) | 19 | 0
Not Completed | 159 | 88
Not completed — Objective Disease Progression | 128 | 30
Not completed — Adverse Event | 18 | 15
Not completed — Withdrawal by Subject | 7 | 10
Not completed — Miscellaneous | 5 | 19
Not completed — Severe Non-compliance to Protocol | 1 | 0
Not completed — Developed Discontinuation Criteria | 0 | 2
Not completed — Withdrew Consent Prior to Dosing | 0 | 12

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are displayed for all participants who started the study. This includes the 12 participants who did not receive treatment in the 'Single Agent Chemotherapy' arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Olaparib 300mg BID | Single Agent Chemotherapy | Total
Number analyzed (Participants) | 178 | 88 | 266
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.5 (9.3) | 60.4 (9.9) | 59.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 88 | 266
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 16 | 47
  Not Hispanic or Latino | 146 | 72 | 218
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 148 | 75 | 223
  Black Or African American | 1 | 1 | 2
  Asian | 24 | 10 | 34
  American Indian Or Alaska Native | 4 | 2 | 6
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: To determine the efficacy of olaparib vs. physician's choice single agent chemotherapy by assessment of Objective Response Rate (ORR) using blinded independent central review (BICR)
  Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria was used by a Blinded Independent Central Review (BICR) to assess participant response to treatment
  ORR is the number of participants with Complete Response (CR) or Partial Response (PR) in the Measurable Disease Analysis Set (MDAS). Complete response is declared when all lesions have disappeared or all lesions have disappeared and all nodal disease is < 10 mm each. Partial response is declared when there is a decrease in sum of diameters of target lesions ≥ 30%.
Time Frame: RECIST follow-up assessments performed every 8 weeks (±1 week), up to 48 weeks, then every 12 weeks (±1 week) from randomisation, assessed from date of first patient randomised to data cut off: 10Oct2018 (approx. 3 years 8 months)
Population: The Measurable Disease Analysis Set (MDAS) includes all participants in the Full Analysis Set (FAS) with measurable disease at baseline (as per RECIST 1.1), determined using Blinded Independent Central Review.
Measure: Number; unit: Count of Participants
Groups:
- Olaparib 300 mg BID: Participants received olaparib twice daily as a 300 mg tablet.
Arm/Group | Olaparib 300 mg BID | Single Agent Chemotherapy
Number analyzed (Participants) | 151 | 72
Count of Participants | 109 | 37
Statistical Analysis 1: Comparison: Olaparib 300 mg BID vs Single Agent Chemotherapy; Test type: Superiority; p = 0.002, Regression, Logistic; Model includes a factor for time to disease progression after the end of last platinum based chemotherapy (6-12 months vs > 12 months); Odds Ratio (OR) = 2.53, 95% CI 2-sided [1.40 to 4.58] — An odds ratio >1 favours the olaparib arm

2. Secondary Outcome: Progression Free Survival (PFS)
Description: To determine the efficacy of single agent olaparib vs. physician's choice single agent chemotherapy by progression free survival (PFS) using BICR assessment according to RECIST 1.1 criteria
  PFS is defined as the time from randomization until the date of objective radiological disease progression according to RECIST 1.1 or death (by any cause in the absence of disease progression) regardless of whether the participant withdrew from randomized therapy or received another anti-cancer therapy prior to disease progression (i.e., date of RECIST progression/death or censoring - date of randomization +1).
Time Frame: as for outcome 1
Population: The Full Analysis Set (FAS) includes all randomized participants and compares the treatment groups on the basis of randomized treatment, regardless of the treatment actually received. Participants who were randomized but did not subsequently go on to receive study treatment were included in the FAS.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg BID | Single Agent Chemotherapy
Number analyzed (Participants) | 178 | 88
Months | 13.4 [10.9 to 14.1] | 9.2 [7.6 to 11.2]
Statistical Analysis 1: Comparison: Olaparib 300 mg BID vs Single Agent Chemotherapy; Test type: Superiority; p = 0.013, Log Rank — Determined using a log-rank test with a factor for time to disease progression after the end of last platinum based chemotherapy (6-12 months vs > 12 months); Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.43 to 0.91] — A hazard ratio < 1 favours the olaparib arm

3. Secondary Outcome: Time From Randomisation to Second Progression (PFS2)
Description: To determine the efficacy of single agent olaparib vs. physician's choice single agent chemotherapy by second progression (PFS2).
  Time from randomization to PFS2 is defined as the time from the date of randomization to the earliest of the progression events subsequent to first progression or death. The date of second progression was recorded by the investigator and defined according to local standard clinical practice, and could involve objective radiological, clinical, cancer antigen-125 (CA-125) progression or death. CA-125 progression was assessed per Gynecological Cancer Intergroup (GCIG) criteria.
Time Frame: Visits to occur every 12 weeks from the date of first progression, assessed from date of first patient randomised to data cut off: 16Apr2021 (approx. 6 years 2 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg BID | Single Agent Chemotherapy
Number analyzed (Participants) | 178 | 88
Months | 23.6 [19.2 to 26.0] | 19.6 [16.9 to 21.8]
Statistical Analysis 1: Comparison: Olaparib 300 mg BID vs Single Agent Chemotherapy; Test type: Superiority; p = 0.229, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.56 to 1.15] — A hazard ratio < 1 favours the olaparib arm

4. Secondary Outcome: Overall Survival (OS)
Description: To determine the efficacy of single agent olaparib vs. physician's choice single agent chemotherapy by overall survival (OS).
  Overall survival is defined as the time from the date of randomisation until death due to any cause.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg BID | Single Agent Chemotherapy
Number analyzed (Participants) | 178 | 88
Months | 34.9 [30.0 to 39.2] | 32.9 [23.5 to 43.2]
Statistical Analysis 1: Comparison: Olaparib 300 mg BID vs Single Agent Chemotherapy; Test type: Superiority; p = 0.714, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.76 to 1.49] — A hazard ratio < 1 favours the olaparib arm

5. Secondary Outcome: Time To Earliest Progression By RECIST 1.1 Or Cancer Antigen (CA) -125 Or Death
Description: To determine the efficacy of single agent olaparib vs. physician's choice single agent chemotherapy by time to earliest progression by RECIST 1.1 or CA-125 or death.
  Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria was used to assess participant response to treatment. CA-125 progression was assessed per Gynecological Cancer Intergroup (GCIG).
Time Frame: RECIST and CA-125 follow-up assessments performed every 8 weeks (±1week), up to 48 weeks, then every 12 weeks (±1week) from randomisation, assessed from date of first patient randomised to data cut off: 10Oct2018 (approx. 3 years 8 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg BID | Single Agent Chemotherapy
Number analyzed (Participants) | 178 | 88
Months | 11.1 [9.7 to 13.8] | 7.9 [6.9 to 9.4]
Statistical Analysis 1: Comparison: Olaparib 300 mg BID vs Single Agent Chemotherapy; Test type: Superiority; p = 0.005, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.41 to 0.85] — A hazard ratio <1 favours the olaparib arm

6. Secondary Outcome: Time From Randomization To First Subsequent Therapy Or Death (TFST)
Description: To determine the efficacy of single agent olaparib vs. physician's choice single agent chemotherapy by time from randomisation to first subsequent therapy or death (TFST)
  TFST is defined as the time from the date of randomisation to the earlier of first subsequent chemotherapy start date or death.
  Anti-cancer treatments include chemotherapy and targeted agents.
Time Frame: Anti-cancer treatments initiated post discontinuation of study treatment and investigator's opinion of response and date of progression recorded, assessed from date of first patient randomised to data cut off: 16Apr2021 (approx. 6 years 2 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg BID | Single Agent Chemotherapy
Number analyzed (Participants) | 178 | 88
Months | 15.4 [13.5 to 17.6] | 10.9 [9.2 to 14.2]
Statistical Analysis 1: Comparison: Olaparib 300 mg BID vs Single Agent Chemotherapy; Test type: Superiority; p < 0.001, Log Rank — Model included factors for number of prior chemotherapy regimens received for ovarian cancer (2 or 3 prior lines vs 4 or more lines) and time to disease progression after the end of last platinum based chemotherapy (6-12 months vs > 12 months); Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.35 to 0.69] — A hazard ratio < 1 favours the olaparib arm

7. Secondary Outcome: Time From Randomization To Second Subsequent Therapy Or Death (TSST)
Description: To determine the efficacy of single agent olaparib vs. physician's choice single agent chemotherapy by time from randomisation to second subsequent therapy or death (TSST)
  TSST was defined as the time from the date of randomisation to the earlier of second subsequent chemotherapy start date or death.
  Anti-cancer treatments include chemotherapy and targeted agents.
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg BID | Single Agent Chemotherapy
Number analyzed (Participants) | 178 | 88
Months | 25.2 [21.3 to 27.8] | 19.9 [18.0 to 24.2]
Statistical Analysis 1: Comparison: Olaparib 300 mg BID vs Single Agent Chemotherapy; Test type: Superiority; p = 0.089, Log Rank — [p-value comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.53 to 1.05] — A hazard ratio < 1 favours the olaparib arm

8. Secondary Outcome: Time From Randomization To Study Treatment Discontinuation Or Death (TDT)
Description: To determine the efficacy of single agent olaparib vs. physician's choice single agent chemotherapy by time to study treatment discontinuation or death (TDT)
  TDT was defined as the time from randomization to the earlier of the date of study treatment discontinuation or death.
Time Frame: Patients randomised to Olaparib administer their tablets orally at a dose of 300 mg twice daily and continue Olaparib until objective disease progression. Assessed from date of first patient randomised to data cut off: 16Apr2021 (approx. 6 years 2 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg BID | Single Agent Chemotherapy
Number analyzed (Participants) | 178 | 88
Months | 13.1 [10.2 to 14.6] | 5.1 [4.7 to 6.5]
Statistical Analysis 1: Comparison: Olaparib 300 mg BID vs Single Agent Chemotherapy; Test type: Superiority; p < 0.001, Log Rank — [p-value comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 0.20, 95% CI 2-sided [0.14 to 0.29] — A hazard ratio < 1 favours the olaparib arm

9. Secondary Outcome: Duration of Response (DoR)
Description: To determine the efficacy of single agent olaparib vs. physician's choice single agent chemotherapy by duration of response (DoR) by BICR using RECIST 1.1 criteria for evaluable patients.
  Duration of response is the time from the first documentation of complete response (CR) or partial response (PR) until the date of progression or death, or the last evaluable RECIST assessment for participants that do not progress or progress after 2 missed assessments. Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria was used to assess participant response to treatment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Olaparib 300 mg BID | Single Agent Chemotherapy
Number analyzed (Participants) | 109 | 37
Months | 9.4 [5.6 to 25.7] | 10.2 [5.5 to 15.3]

10. Secondary Outcome: Time to Response (TTR)
Description: To determine the efficacy of single agent olaparib vs. physician's choice single agent chemotherapy by time to response (TTR) by BICR using RECIST 1.1 criteria for evaluable patients.
  TTR was defined as the time from randomization until the date of first documented response by Blinded independent central review (BICR) assessment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Olaparib 300 mg BID | Single Agent Chemotherapy
Number analyzed (Participants) | 109 | 37
Months | 2.0 [1.8 to 3.9] | 3.5 [1.8 to 3.7]

11. Secondary Outcome: Mean Change From Baseline In Trial Outcome Index (TOI) Score
Description: To compare the efficacy of single agent olaparib versus physician's choice single agent chemotherapy on the Health-related Quality of Life (HRQoL) as measured by the trial outcome index (TOI) of the Functional Assessment of Cancer Therapy - Ovarian (FACT-O)
  The TOI score was derived from the sum of the scores of the 25 items included in the physical well-being (7 items), functional well-being (7 items), and additional concerns ovarian cancer subscale (11 items) of the FACT-O questionnaire Version 4. TOI score ranges from 0 to 100, a higher score indicates a higher HRQoL. A negative change in score from baseline indicated a worsening in symptoms.
Time Frame: Baseline (Day 1) to Week 48 (±1 week). DCO: 10Oct2018
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Selected Chemotherapy: Participants received physician's choice of chemotherapy, out of weekly paclitaxel, topotecan, pegylated liposomal doxorubicin, or gemcitabine.
Arm/Group | Olaparib 300 mg BID | Selected Chemotherapy
Number analyzed (Participants) | 167 | 62
Scores on a scale | -2.4 (11.1) | -3.6 (9.8)
Statistical Analysis 1: Comparison: Olaparib 300 mg BID vs Selected Chemotherapy; Test type: Superiority; p = 0.108, Mixed Models Analysis; Model includes factors for patient, treatment, visit, treatment by visit interaction, baseline TOI score and baseline TOI score by visit interaction; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [-0.5 to 5.5]

12. Secondary Outcome: Number of Participants Who Show an Improvement in TOI Score
Description: To compare the efficacy of single agent olaparib versus physician's choice single agent chemotherapy on the Health-related Quality of Life (HRQoL) as measured by the trial outcome index (TOI) of the Functional Assessment of Cancer Therapy - Ovarian (FACT-O)
  The TOI score was derived from the sum of the scores of the 25 items included in the physical well-being (7 items), functional well-being (7 items), and additional concerns ovarian cancer subscale (11 items) of the FACT-O questionnaire Version 4. TOI score ranges from 0 to 100, a higher score indicates a higher health-related quality of life (HRQoL). A change in at least 10 points was considered clinically relevant.
Time Frame: Baseline (Day 1) to Week 48 (±1 week). DCO: 10Oct2018
Population: as for outcome 2
Measure: Number; unit: Count of Participants
Arm/Group | Olaparib 300 mg BID | Single Agent Chemotherapy
Number analyzed (Participants) | 168 | 69
Count of Participants | 25 | 5
Statistical Analysis 1: Comparison: Olaparib 300 mg BID vs Single Agent Chemotherapy; Test type: Superiority; p = 0.092, Regression, Logistic — Estimated from an unadjusted logistic regression model; Odds Ratio (OR) = 2.24, 95% CI 2-sided [0.88 to 6.86] — An odds ratio > 1 favours the olaparib arm

13. Secondary Outcome: Objective Response Rate (ORR) in Breast Cancer Susceptibility (BRCA) Gene Population by Blinded Independent Central Review (BICR)
Description: BRCA gene population includes participants identified as having a deleterious or suspected deleterious variant in either of the BRCA genes using variants identified with current and future BRCA mutation assays (eg, gene sequencing and large rearrangement analysis).
  The number of participants with complete or partial response per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria. Partial response is declared when there is a decrease in sum of target disease ≥ 30%. Complete response is declared when all lesions have disappeared or all lesions have disappeared and all nodal disease is < 10 mm each.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Count of Participants
Arm/Group | Olaparib 300 mg BID | Single Agent Chemotherapy
Number analyzed (Participants) | 144 | 70
Count of Participants | 103 | 36
Statistical Analysis 1: Comparison: Olaparib 300 mg BID vs Single Agent Chemotherapy; Test type: Superiority; p = 0.004, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.40, 95% CI 2-sided [1.32 to 4.39] — An odds ratio > 1 favours the olaparib arm

14. Secondary Outcome: Number of Participants Who Experienced Disease Progression or Death in BRCA Gene Population by Blinded Independent Central Review (BICR)
Description: BRCA gene population includes participants identified as having a deleterious or suspected deleterious variant in either of the BRCA genes using variants identified with current and future BRCA mutation assays (eg, gene sequencing and large rearrangement analysis).
  Progressive disease was defined as at least 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: Count of Participants
Arm/Group | Olaparib 300 mg BID | Single Agent Chemotherapy
Number analyzed (Participants) | 170 | 84
Count of Participants | 105 | 48
Statistical Analysis 1: Comparison: Olaparib 300 mg BID vs Single Agent Chemotherapy; Test type: Superiority; p = 0.014, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.42 to 0.91] — A hazard ratio < 1 favours the olaparib arm

15. Secondary Outcome: Number of Participants Who Experienced Second Progression or Death (PFS2) in BRCA Gene Population
Description: BRCA gene population includes participants identified as having a deleterious or suspected deleterious variant in either of the BRCA genes using variants identified with current and future BRCA mutation assays (eg, gene sequencing and large rearrangement analysis).
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number; unit: Count of Participants
Arm/Group | Olaparib 300 mg BID | Single Agent Chemotherapy
Number analyzed (Participants) | 170 | 84
Count of Participants | 110 | 48
Statistical Analysis 1: Comparison: Olaparib 300 mg BID vs Single Agent Chemotherapy; Test type: Superiority; p = 0.213, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.56 to 1.14] — A hazard ratio < 1 favours the olaparib arm

16. Secondary Outcome: Overall Survival (OS) in BRCA Gene Population
Description: BRCA gene population includes participants identified as having a deleterious or suspected deleterious variant in either of the BRCA genes using variants identified with current and future BRCA mutation assays (eg, gene sequencing and large rearrangement analysis).
  OS in BRCA gene population was measured by the number of participants who died due to any cause.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number; unit: Count of Participants
Arm/Group | Olaparib 300 mg BID | Single Agent Chemotherapy
Number analyzed (Participants) | 170 | 84
Count of Participants | 111 | 45
Statistical Analysis 1: Comparison: Olaparib 300 mg BID vs Single Agent Chemotherapy; Test type: Superiority; p = 0.699, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.76 to 1.51] — A hazard ratio < 1 favours the olaparib arm

17. Secondary Outcome: Number of Participants Who Discontinued Study Treatment or Died in BRCA Gene Population
Description: as for outcome 15
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Number; unit: Count of Participants
Arm/Group | Olaparib 300 mg BID | Single Agent Chemotherapy
Number analyzed (Participants) | 170 | 84
Count of Participants | 151 | 76
Statistical Analysis 1: Comparison: Olaparib 300 mg BID vs Single Agent Chemotherapy; Test type: Superiority; p < 0.001, Log Rank — [p-value comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 0.18, 95% CI 2-sided [0.12 to 0.27] — A hazard ratio < 1 favours the olaparib arm

18. Secondary Outcome: Number of Participants Who Received Subsequent Chemotherapy or Died in BRCA Gene Population
Description: BRCA gene population includes participants identified as having a deleterious or suspected deleterious variant in either of the BRCA genes using variants identified with current and future BRCA mutation assays (eg, gene sequencing and large rearrangement analysis).
  Anti-cancer treatments include chemotherapy and targeted agents.
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Number; unit: Count of Participants
Arm/Group | Olaparib 300 mg BID | Selected Chemotherapy
Number analyzed (Participants) | 170 | 84
Count of Participants | 138 | 66
Statistical Analysis 1: Comparison: Olaparib 300 mg BID vs Selected Chemotherapy; Test type: Superiority; p < 0.001, Log Rank — [p-value comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.33 to 0.66] — A hazard ratio < 1 favours the olaparib arm

19. Secondary Outcome: Number of Participants Who Received Second Subsequent Chemotherapy or Died in BRCA Gene Population
Description: as for outcome 18
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Number; unit: Count of Participants
Arm/Group | Olaparib 300 mg BID | Single Agent Chemotherapy
Number analyzed (Participants) | 170 | 84
Count of Participants | 127 | 56
Statistical Analysis 1: Comparison: Olaparib 300 mg BID vs Single Agent Chemotherapy; Test type: Superiority; p = 0.055, Log Rank — [p-value comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.51 to 1.01] — A hazard ratio < 1 favours the olaparib arm

20. Secondary Outcome: Geometric Mean Plasma Concentration of Olaparib
Description: Summary of plasma concentrations (ug/mL) of olaparib
Time Frame: Day 1, 1 hour post-dose and Day 29 pre-dose. DCO: 10Oct2018
Population: The pharmacokinetic (PK) analysis set includes all participants who received an olaparib dose and provided evaluable plasma concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Olaparib 300 mg BID
Number analyzed (Participants) | 66
μg/mL
  Day 1, 1 hour post-dose | 4.76 (112.93)
  Day 29, pre-dose: number analyzed (Participants) | 42
  Day 29, pre-dose | 1.78 (100.54)

21. Secondary Outcome: Number of Participants Who Experience at Least One Adverse Event (AE)
Description: An AE is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product.
Time Frame: Safety Follow-up 30 days after last dose of IP, assessed from the date of first patient randomised to data cut off: 16Apr2021 (approx. 6 years 2 months)
Population: The safety analysis set includes all participants who received at least 1 dose of randomized study treatment, olaparib or chemotherapy.
Measure: Number; unit: Count of Participants
Arm/Group | Olaparib 300 mg BID | Single Agent Chemotherapy
Number analyzed (Participants) | 178 | 76
Count of Participants | 175 | 73

ADVERSE EVENTS:
Time Frame: Includes all AEs that had a start date or a worsening (increase in CTCAE grade) after the start of treatment up until the end of the 30 day follow-up period. The 30 day follow-up period will be defined as 30 days following discontinuation of olaparib/chemotherapy treatment. Assessed from randomisation to data cut off. DCO: 16Apr2021
Description: All-Cause Mortality was collected for the Full Analysis Set (FAS).
  Serious Adverse Events and Other Adverse Events were collected for the Safety Analysis Set (SAS), which includes patients who received at least 1 dose of the randomised study treatment.
Groups:
- Olaparib 300 mg bd: Participants received olaparib twice daily as a 300 mg tablet.
Arm/Group | Olaparib 300 mg bd | Single Agent Chemotherapy
All-Cause Mortality (participants affected / at risk) | 116/178 | 46/88
Serious Adverse Events (participants affected / at risk) | 46/178 | 14/76
Other Adverse Events (participants affected / at risk) | 173/178 | 73/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 300 mg bd (N=178) | Single Agent Chemotherapy (N=76)
Anaemia (Blood and lymphatic system disorders) | 6 (7) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Corneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3)
Asthenia (General disorders) | 2 (2) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 300 mg bd (N=178) | Single Agent Chemotherapy (N=76)
Anaemia (Blood and lymphatic system disorders) | 87 (163) | 19 (22)
Neutropenia (Blood and lymphatic system disorders) | 29 (41) | 22 (37)
Abdominal distension (Gastrointestinal disorders) | 11 (12) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 16 (19) | 8 (9)
Alanine aminotransferase increased (Investigations) | 5 (7) | 4 (4)
Neutrophil count decreased (Investigations) | 16 (34) | 10 (36)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (28) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 5 (6) | 8 (8)
Depression (Psychiatric disorders) | 9 (9) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 27 (42)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (8) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 13 (17) | 9 (14)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 41 (80) | 11 (15)
Abdominal pain upper (Gastrointestinal disorders) | 21 (36) | 4 (4)
Constipation (Gastrointestinal disorders) | 24 (28) | 17 (23)
Diarrhoea (Gastrointestinal disorders) | 52 (149) | 13 (16)
Dyspepsia (Gastrointestinal disorders) | 19 (26) | 7 (8)
Flatulence (Gastrointestinal disorders) | 1 (1) | 4 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 (10) | 2 (2)
Nausea (Gastrointestinal disorders) | 115 (240) | 24 (47)
Stomatitis (Gastrointestinal disorders) | 8 (11) | 14 (28)
Vomiting (Gastrointestinal disorders) | 66 (165) | 14 (20)
Asthenia (General disorders) | 35 (52) | 12 (16)
Leukopenia (Blood and lymphatic system disorders) | 13 (24) | 6 (6)
Fatigue (General disorders) | 66 (91) | 20 (26)
Influenza like illness (General disorders) | 7 (8) | 4 (5)
Mucosal inflammation (General disorders) | 5 (5) | 10 (11)
Oedema peripheral (General disorders) | 16 (24) | 10 (16)
Pyrexia (General disorders) | 21 (28) | 8 (10)
Bronchitis (Infections and infestations) | 10 (12) | 2 (2)
Urinary tract infection (Infections and infestations) | 21 (26) | 4 (4)
Blood creatinine increased (Investigations) | 14 (25) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 6 (8) | 4 (4)
White blood cell count decreased (Investigations) | 18 (34) | 9 (22)
Decreased appetite (Metabolism and nutrition disorders) | 26 (30) | 9 (9)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 (13) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (16) | 3 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 (19) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (20) | 6 (11)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (14) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (35) | 6 (10)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 (21) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (18) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (13) | 6 (7)
Dizziness (Nervous system disorders) | 25 (65) | 6 (6)
Dysgeusia (Nervous system disorders) | 13 (16) | 6 (6)
Headache (Nervous system disorders) | 29 (79) | 9 (11)
Paraesthesia (Nervous system disorders) | 7 (8) | 5 (6)
Anxiety (Psychiatric disorders) | 4 (6) | 6 (6)
Insomnia (Psychiatric disorders) | 17 (18) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (24) | 10 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 (26) | 8 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (11) | 12 (12)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT02282020/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT02282020/SAP_001.pdf